CLINICAL TRIAL: NCT06441981
Title: Closing the Gap in Public Perception and Policy for SARS-CoV-2 Whole Genome Sequencing and Genomics for All
Brief Title: Public Perception and Policy for SARS-CoV-2 Whole Genome Sequencing and Genomics for All
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Collaborators: Oxford University Clinical Research Unit (Unknown)
Responsible Party: Principal Investigator, Rina Agustina, Principal Investigator, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: WGS Project
Record Dates: First submitted 2024-05-31; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Knowledge, Attitudes, Practice
Keywords: Genome Sequencing; Public Perception; Public Policy; COVID-19
MeSH Terms: conditions — Behavior; COVID-19 | interventions — Educational Status

STUDY DESIGN:
Intervention Model Description: The questionnaire in whatsapp chatbot format will be given to 100 and up to 200 persons from each targeted population. There Four targeted population namely, The public overall (comprised mostly of 18-29 years old adults whom have the most cases), Vulnerable groups (including the elderly between 50-80 years old, parents of children 0-12 years, and pregnant women), Doctors and other frontline health workers, and Program implementers and policy makers.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral Education (Other): Educational material is provided via WhatsApp chatbot. After being educated, respondents were given a test to determine the increase in understanding of the material.
  Interventions: Behavioral: Education

INTERVENTIONS:
Behavioral: Education — Educational material brochures will be given to 800 respondents. Educational material is provided via WhatsApp chatbot. After being educated, respondents were given a test to determine the increase in understanding of the material.

SUMMARY:
Gap in understanding undermines government and public support for SC2-WGS, and other wide-scale genomic sequencing (Gut microbiome, Genome Wide Sequencing for Prenatal Detection, Tuberculosis Metagenomic sequencing, Nutrigenetics and Cancer Next Generation Sequencing) as a routine part of the pandemic response, especially in low- and middle-income countries. However, such gaps can be closed with systematic efforts to define and measure specific misperceptions, and subsequently design and use targeted messages and promotional materials. We propose here in the following specific aims to first determine the entire set of beliefs and emotions regarding SC2-WGS and other genomic sequencing (Gut microbiome, Genome Wide Sequencing for Prenatal Detection, Tuberculosis Metagenomic sequencing, Nutrigenetics and Cancer Next Generation Sequencing), then identify and measure limiting belief constructs, and then create social media and communication media to address and overcome limiting beliefs strategically. The goal is to increase public and policymaker support for SC2-WGS and other genomic sequencing (Gut microbiome, Genome Wide Sequencing for Prenatal Detection, Tuberculosis Metagenomic sequencing, Nutrigenetics and Cancer Next Generation Sequencing) resources and actions for pandemic control.

DETAILED DESCRIPTION:
Implementing WGS, it is advisable to involve a variety of relevant actors and to consider the opinions of various stakeholders, including those who are not professionals in the field. This might resolve the implementation problem that could occur if psychological and social dimensions or, in other words, not strictly scientific criteria are not adequately integrated in decision making concerning complex issues such as innovations in genetics. In most cases, the reaction towards genetic information corresponds with a specific personal view of how to handle medical information and thus amplifies already existing mental phenomena (fear, stress, worries, etc.), tendencies of self-improvement and self-care and curiosity and playfulness.38 In the Study from Lewis et al, investigated in this relation the specific personality traits of participants of the first implementations of WGS, who were characterized as optimistic and resilient. This is a phenomenon often found in the group of early adopters of new technologies in general as described in the dimension knowing as empowerment to act, for some people, the willingness to know is caused by an attitude of openness towards the unknown and the desire to open new scenarios that could activate new opportunities for research as well as for themselves. This perspective highly reflects the currently dominant societal goal of health prevention and the main health policy discourse and practice of precaution. People have different perceptions of WGS and its imaginable integration into our health care system or our daily lives, and various approaches to decision-making regarding the potential use of WGS could be observed.

There are suboptimal national resources, inadequate specimen sampling strategies, to optimize epidemiological and clinical inference. There is a gap in the meta-data to interpret SC2-WGS information and other genomic sequencing (Gut microbiome, Genome Wide Sequencing for Prenatal Detection, Tuberculosis Metagenomic sequencing, Nutrigenetics and Cancer Next Generation Sequencing) in a complete and rapid manner. This understanding gap can undermine broad-scale government and public support as a routine part of the pandemic response, especially in low- and middle-income countries.

Therefore an intervention is needed in the form of genomic sequencing education. Before the intervention stage, there will be taking survey data which will be collected using the themes from the FGD results and will focus on assessing public perceptions regarding SC2-WGS and other genomic sequencing. These themes will be formulated into short statements and answered by respondents using a Likert scale. The survey will involve 100-200 respondents via WhatsApp chat bot. Subjects will be asked to express their reactions to short statements on a 4-point Likert scale. The subject will also be asked to express his emotional reaction to the statement with a series of binary questions related to positive or negative feelings. The survey results will be analyzed quantitatively to see the total score and distribution of each statement.

The next stage in this research is to develop social media and communication media. At this stage we will formulate public messages and strategies to improve perceptions based on the survey results. The public message formulated will be useful for educating the public using various social media platforms.

The intervention stage will be carried out by distributing information regarding genome sequencing via bots. After the intervention is carried out, changes in perception will be assessed before and after the intervention through pre-test and post-test questionnaires

ELIGIBILITY:
Inclusion Criteria:

* Living or working in Jakarta
* Young adult
* Adult
* Elderly
* Health workers
* Public Policy

Exclusion Criteria:

- Living or working outside Jakarta

Ages: 21 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-10-31 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Knowledge | 2 months
  Assessment of respondents' knowledge regarding the educational material provided, calculated based on the number of questions answered correctly.

CONTACTS AND LOCATIONS:
Overall Officials: Rina Agustina, Principal Investigator — https://imeri.fk.ui.ac.id
Locations (1):
- Department of Nutrition (FKUI-RSCM); and Human Nutrition Research Center, Indonesian Medical Education Research Institute (HNRC-IMERI) Faculty of Medicine, Universitas Indonesia, Jakarta Pusat, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Schumann S, Gschmeidler B, Pellegrini G. Knowing, relationships and trust-citizens' perceptions of whole genome sequencing for the Genetics Clinic of the Future. J Community Genet. 2021 Jan;12(1):67-80. doi: 10.1007/s12687-020-00486-0. Epub 2020 Sep 30. PMID 32997319
- [Background] Lewis KL, Han PK, Hooker GW, Klein WM, Biesecker LG, Biesecker BB. Characterizing Participants in the ClinSeq Genome Sequencing Cohort as Early Adopters of a New Health Technology. PLoS One. 2015 Jul 17;10(7):e0132690. doi: 10.1371/journal.pone.0132690. eCollection 2015. PMID 26186621
- See also: Re-Thinking Science: Knowledge and the Public in an Age of Uncertainty — https://www.academia.edu/17329773/Re_Thinking_Science_Knowledge_and_the_Public_in_an_Age_of_Uncertainty_by_Helga_Nowotny_Peter_Scott_and_Michael_Gibbons